CLINICAL TRIAL: NCT00002101
Title: A Three-Arm Comparative Trial for the Treatment of MAC Bacteremia in AIDS: A Clarithromycin/Ethambutol Regimen Containing Rifabutin (450 Mg) or Rifabutin (300 Mg) or Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacia (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 048D; CS 087250-999
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: Rifabutin; Mycobacterium avium-intracellulare Infection; Drug Therapy, Combination; Ethambutol; Acquired Immunodeficiency Syndrome; Clarithromycin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ethambutol; Clarithromycin; Rifabutin

INTERVENTIONS:
Drug: Ethambutol hydrochloride
Drug: Clarithromycin
Drug: Rifabutin

SUMMARY:
To compare the efficacy of clarithromycin/ethambutol with placebo or with rifabutin at two different doses in reducing colony-forming units (CFUs) by 2 or more logarithms in patients with Mycobacterium avium Complex bacteremia and maintaining this response until 16 weeks post-randomization. To assess survival and comparative tolerability among the three treatment regimens.

DETAILED DESCRIPTION:
Patients are randomized to receive clarithromycin and ethambutol plus either placebo or rifabutin at one of two doses. Treatment continues indefinitely. AS PER AMENDMENT 04/19/94: Doses of rifabutin have been lowered.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Isoniazid for TB prophylaxis ONLY.

Patients must have:

* HIV infection.
* MAC infection.
* Life expectancy of at least 16 weeks.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Perceived unreliability or unavailability for frequent monitoring.

Concurrent Medication:

Excluded:

* Antimycobacterial drugs other than the study drugs.
* Carbamazepine.
* Terfenadine.
* Theophylline.

Patients with the following prior condition are excluded:

History of hypersensitivity to rifabutin, rifampin, erythromycin, clarithromycin, azithromycin, or ethambutol.

Prior Medication:

Excluded within 7 days prior to study entry:

* Rifabutin.
* Rifampin.
* Ethionamide.
* Cycloserine.
* Clofazimine.
* Ethambutol.
* Amikacin.
* Ciprofloxacin.
* Ofloxacin.
* Sparfloxacin.
* Azithromycin.
* Clarithromycin.
* Pyrazinamide.

Excluded within 14 days prior to study entry:

* Carbamazepine.
* Terfenadine.
* Theophylline.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - McDowell Clinic, Phoenix, Arizona
  - Maricopa Med Research Foundation, Phoenix, Arizona
  - Bay Harbor Hosp, Harbor City, California
  - Ctr for Special Immunology, Irvine, California
  - Combat Group, Los Angeles, California
  - Cedars Sinai Med Ctr, Los Angeles, California
  - Highland Gen Hosp / San Francisco Gen Hosp, Oakland, California
  - HIV Research Group, San Diego, California
  - UCSD / Ctr for Special Immunology, San Diego, California
  - Saint Francis Mem Hosp, San Francisco, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Sunnyvale Med Clinic, Sunnyvale, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr, Washington D.C., District of Columbia
  - Infectious Disease Consultants, Altamonte Springs, Florida
  - TheraFirst Med Ctrs Inc, Fort Lauderdale, Florida
  - Dr Frank Tornaka, Fort Lauderdale, Florida
  - Gary Richmond MD, Fort Lauderdale, Florida
  - Dr Nelson Zide, Hollywood, Florida
  - Ctr for Special Immunology, Miami Beach, Florida
  - Dr Barry Rodwick, Safety Harbor, Florida
  - Bay Area AIDS Consortium, Tampa, Florida
  - Infectious Disease Research Consortium of Georgia, Atlanta, Georgia
  - Dr Daniel Berger, Chicago, Illinois
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Tulane Univ Med School, New Orleans, Louisiana
  - Dr Arnold Markowitz, Keego Harbor, Michigan
  - Univ of Nebraska Med Ctr / HIV Clinic, Omaha, Nebraska
  - East Orange Veterans Administration Med Ctr, East Orange, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Long Island Jewish Med Ctr, New Hyde Park, New York
  - Chelsea Village Med Ctr / Saint Vincent's Hosp, New York, New York
  - Community Health Network, Rochester, New York
  - Nalle Clinic, Charlotte, North Carolina
  - Polyclinic Med Ctr, Harrisburg, Pennsylvania
  - Buckley Braffman Stern Med Associates, Philadelphia, Pennsylvania
  - Charleston Veterans Administration Med Ctr, Charleston, South Carolina
  - Dr Alfred F Burnside Jr, Columbia, South Carolina
  - Central Texas Med Foundation, Austin, Texas
  - Houston Veterans Administration Med Ctr, Houston, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Univ of Wisconsin School of Medicine, Madison, Wisconsin
  - Milwaukee County Med Complex, Milwaukee, Wisconsin